CLINICAL TRIAL: NCT04567693
Title: Reducing Time to Spaced-out Appointments for Newly-diagnosed People Living With HIV: a Pilot Study
Brief Title: Reducing Time to Spaced-out Appointments for Newly-diagnosed People Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Albert Einstein College of Medicine (Other); Rwanda Military Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-11551; K23MH114752 (NIH)
Record Dates: First submitted 2020-09-17; First posted 2020-09-28 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Hiv; Aids
Keywords: Rwanda; Treat All; Antiretroviral therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early 1 (Experimental): Advance to spaced-out appointments at month 6 after a single viral load is measured.
  Interventions: Other: Early spaced-out appointments
- Early 2 (Experimental): Advance to spaced-out appointments at month 6 after two viral loads are measured.
  Interventions: Other: Early spaced-out appointments
- Usual Care (No Intervention): Do not advance to spaced-out appointments during study period

INTERVENTIONS:
Other: Early spaced-out appointments — Newly-diagnosed PLWH currently attend health centers monthly for ART pick-up and quarterly for clinical visits. In the intervention arms, participants will attend health centers quarterly for ART pick-up and semi-annually for clinical visits.
  Arms: Early 1; Early 2

SUMMARY:
The objectives of this study are to pilot test the effect of reducing time to spaced-out appointments from 18 to 6 months for newly-diagnosed people living with HIV (PLWH) in Rwanda who have initiated antiretroviral therapy (ART). PLWH are currently required to visit the health center monthly for ART and clinical appointments for the first 18 months on ART, after which they can attend quarterly. Reducing the time to spaced-out appointments from 18 to 6 months has the potential to reduce the burden on patients and the health system, but may lead to suboptimal treatment outcomes. To better understand the effects of early spaced-out appointments as well as the degree of viral load monitoring needed to determine stability on ART, the investigators will conduct a 3-arm pilot intervention study. The investigators will randomize participants to 1) 6-month advancement to spaced-out appointments after 1 viral load measurement; 2) 6-month advancement to spaced-out appointments after 2 viral load measurements; or 3) usual care. The investigators will compare the study arms with respect to viral suppression at 12 months after enrollment in ART care (primary outcome) and appointment/ pharmacy adherence (secondary outcome).

DETAILED DESCRIPTION:
Most countries in sub-Saharan Africa have adopted differentiated care models for people living with HIV (PLWH), including Rwanda. Current Rwandan HIV guidelines classify newly-diagnosed PLWH as "unstable", requiring monthly visits to the health facility. Before they can advance to being "stable" patients, with spaced-out appointments that allow them to visit the health facility every three months, they must be on antiretroviral therapy (ART) for 18 months and virally suppressed on two consecutive measurements. Patients face multiple barriers to attending frequent appointments including structural issues (such as distance to the health facility, transportation cost, long waiting times) and facing stigma while traveling to and while at the health facility. Reducing the time newly-diagnosed PLWH spend in the "unstable" category could potentially decrease the burden on patients and the health facility and potentially decrease the costs of frequent appointments. The investigators therefore propose a pilot study to examine the effect of reducing the time from ART initiation to advancement to the "stable" category from 18 to 6 months. The investigators will enroll 90 patients: 30 will be randomized to 6-month advancement to spaced out appointments after 1 viral load is measured (at 5 months after enrollment in ART care) ("Early 1"); 30 will be randomized to 6-month advancement to spaced-out appointments after 2 viral loads are measured (at 3- and 5-months after enrollment in ART care) ("Early 2"); and 30 will be randomized to continue in usual care with monthly visits ("Usual care"). The investigators will compare study arms with respect to viral suppression at 12 months (primary outcome) and appointment/pharmacy adherence (secondary outcome). The investigators hypothesize that reducing the time to the "stable" category with spaced out appointments will be feasible, acceptable, not inferior to 18 months with respect to viral suppression or adherence, and will be cost-effective.

ELIGIBILITY:
Inclusion Criteria:

1. ≥15 years;
2. newly-diagnosed with HIV (within 6 months);
3. enrolled in care at study health facility;
4. initiated ART.

Exclusion Criteria:

1. planning on moving away from health center/Kigali in the next 12 months;
2. unable to provide informed consent;
3. enrolled in care while pregnant;
4. co-infected with tuberculosis;
5. concurrent known mental health or substance use disorder.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ross, Principal Investigator — Montefiore Medical Center
Locations (1):
- Rwanda Military Hospital, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study, we have elected to not allow for data to be available to other researchers for secondary analyses.

REFERENCES:
- [Derived] Ross J, Anastos K, Hill S, Remera E, Rwibasira GN, Ingabire C, Umwiza F, Munyaneza A, Muhoza B, Zhang C, Nash D, Yotebieng M, Murenzi G. Reducing time to differentiated service delivery for newly-diagnosed people living with HIV in Kigali, Rwanda: a pilot, unblinded, randomized controlled trial. BMC Health Serv Res. 2024 Apr 30;24(1):555. doi: 10.1186/s12913-024-10950-z. PMID 38693537
- [Derived] Ross J, Murenzi G, Hill S, Remera E, Ingabire C, Umwiza F, Munyaneza A, Muhoza B, Habimana DS, Mugwaneza P, Zhang C, Yotebieng M, Anastos K. Reducing time to differentiated service delivery for newly diagnosed people living with HIV in Kigali, Rwanda: study protocol for a pilot, unblinded, randomised controlled study. BMJ Open. 2021 Apr 24;11(4):e047443. doi: 10.1136/bmjopen-2020-047443. PMID 33895720

RESULTS

PARTICIPANT FLOW:
Groups:
- Early 1: Advance to spaced-out appointments at month 6 after a single viral load is measured.
  Early spaced-out appointments: Newly-diagnosed PLWH currently attend health centers monthly for ART pick-up and quarterly for clinical visits. In this arm, starting at 6 months after ART initiation, participants whose 5-month viral load are suppressed attend health centers quarterly for ART pick-up and semi-annually for clinical visits.
- Early 2: Advance to spaced-out appointments at month 6 after two viral loads are measured.
  Early spaced-out appointments: Newly-diagnosed PLWH currently attend health centers monthly for ART pick-up and quarterly for clinical visits. In this arm, starting at 6 months after ART initiation, participants whose 3- and 5-month viral loads are both suppressed attend health centers quarterly for ART pick-up and semi-annually for clinical visits.
Period: Overall Study
Arm/Group | Early 1 | Early 2 | Usual Care
Started | 32 | 31 | 30
Completed | 30 | 31 | 24
Not Completed | 2 | 0 | 6
Not completed — Death | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Withdrawal by investigative team (participants did not meet eligibility criteria) | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: 3 enrolled participants were assigned to groups (one participant to the 'Early 1' group and two participants to the 'Usual Care' group), but subsequently withdrawn from the study when it became clear that they did not meet eligibility criteria. Their data were not included in baseline analysis or any further analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early 1 | Early 2 | Usual Care | Total
Number analyzed (Participants) | 31 | 31 | 28 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (10) | 33 (13) | 29 (6) | 31 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 20 | 60
  Male | 11 | 11 | 8 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Rwanda | 31 | 31 | 28 | 90
ART Adherence [Mean (Standard Deviation); unit: Days of ART missed in last 30 days] — Days of ART missed in last 30 days
  Days of ART missed in last 30 days | 0.1 (0.72) | 0.03 (0.18) | 0.04 (0.19) | 0.06 (0.44)
Satisfaction with care [Mean (Standard Deviation); unit: units on a scale] — The Satisfaction With Care scale is a 9-item scale containing questions about satisfaction with clinical (n=6) and non-clinical elements (n=3) of health care. Participants describe satisfaction with each element on a 5-point Likert scale (very unsatisfied [1], not satisfied [2], no opinion [3], satisfied [4], very satisfied [5]). Satisfaction with clinical and non-clinical care elements are reported separately, by summing scores (1-5) for each item and then dividing by the number of items within each subscale. Subscale scores range from 1 to 5; higher scores indicate greater satisfaction.
  units on a scale
    Non-clinical | 4.15 (0.34) | 4.12 (0.34) | 4.11 (0.49) | 4.13 (0.40)
    Clinical | 3.81 (0.28) | 3.84 (0.21) | 3.85 (0.24) | 3.83 (0.24)
Enacted and Internalized Stigma [Mean (Standard Deviation); unit: units on a scale] — As measured by the HIV/AIDS Stigma Instrument-PLWA (HASI-P) Scale. The HASI-P is a 33-item scale that contains questions in 6 different stigma-related domains or factors. For each item, participants are asked to describe the frequency of experienced stigmatizing events in the past 3 months on a 4-point Likert scale (0- Never, 1- Once or twice, 2- Several times, or 3- Most of the time), with higher scores indicating greater stigma. The instrument is scored by summing the scores (0-3) for each item and then dividing by the number of items within each factor (enacted or internalized stigma).
  units on a scale
    Enacted | 1.04 (0.20) | 1.03 (0.09) | 1.00 (0.01) | 1.00 (0.11)
    Internalized | 2.02 (0.77) | 1.62 (0.72) | 2.08 (0.97) | 1.90 (0.80)
Quality of life [Mean (Standard Deviation); unit: units on a scale] — Repeated measures analysis of participant quality of life as measured by the EuroQOL-5 Dimension-5 Levels (EQ-5D-5L) Visual Analog Scale (VAS). The EQ-5D-5L is a 5-level scale that measures self-rated problems (no problems, slight problems, moderate problems, severe problems and extreme problems) in 5 domains (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) as well as self-rated health. For this measure, we chose to use only the VAS, which asks respondents to rate their overall health from 0-100, with higher scores indicating greater self-rated health.
  units on a scale | 45.0 (14.0) | 45.5 (17.7) | 37.9 (16.2) | 42.9 (16.2)
Anticipated stigma [Mean (Standard Deviation); unit: units on a scale] — As measured by an adapted version of the HIV stigma scale (anticipated stigma). Anticipated stigma is rated on a 5-point Likert-type scale (Very Unlikely [1] to Very Likely [5]), with higher scores indicating greater stigma. Items are averaged to create a composite score.
  units on a scale | 2.40 (.074) | 2.40 (0.72) | 2.43 (0.85) | 2.40 (0.70)

OUTCOME MEASURES:

1. Primary Outcome: Viral Suppression
Description: Percentage of participants with suppressed viral load (less than 200 copies/ml)
Time Frame: Measured at 12 months after enrollment into ART care
Population: Note: as the primary, intention to treat outcome, persons who did not complete the study were treated as being not virally suppressed. 3 enrolled participants were assigned to groups (one participant to the 'Early 1' group and two participants to the 'Usual Care' group), but subsequently withdrawn from the study when it became clear that they did not meet eligibility criteria. Their data were not included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 31 | 31 | 28
Participants | 25 | 25 | 19

2. Secondary Outcome: Appointment Adherence
Description: Proportion of participants that attended all pharmacy and clinical appointments
Time Frame: Measured at 12 months after enrollment into ART care
Population: Appointment adherence was defined in the protocol as the proportion of participants in each arm who attended all scheduled clinical appointments and ART pick-ups during the study. We planned to ascertain appointment adherence through review of participants' medical files at the conclusion of the study. During medical file review, it became apparent that scheduled appointments (i.e. next planned) were inconsistently documented. We therefore were unable to accurately ascertain this outcome.
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Participant Acceptability of Reduced Time to Spaced-out Appointments
Description: The Satisfaction With Care scale is a 9-item scale containing questions about satisfaction with clinical (n=6) and non-clinical elements (n=3) of health care. Participants describe satisfaction with each element on a 5-point Likert scale (very unsatisfied [1], not satisfied [2], no opinion [3], satisfied [4], very satisfied [5]). Satisfaction with clinical and non-clinical care elements are reported separately, by summing scores (1-5) for each item and then dividing by the number of items within each subscale. Subscale scores range from 1 to 5; higher scores indicate greater satisfaction.
Time Frame: Measured at 12 months after enrollment into ART care
Measure: Mean (Standard Deviation); unit: score on a scale (Likert)
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 30 | 31 | 24
score on a scale (Likert)
  Non-clinical | 4.2 (0.5) | 4.3 (0.5) | 4.2 (0.6)
  Clinical aspects of care | 3.9 (0.3) | 4.0 (0.3) | 3.9 (0.3)

4. Secondary Outcome: Provider Acceptability of Reduced Time to Spaced-out Appointments
Description: Acceptability of reduced time to spaced-out appointments, as measured by the number of instances when providers overrode the study assignment. Override could only occur a maximum of one time for each participant.
Time Frame: Measured at 12 months after enrollment into ART care
Population: Overriding of study assignment was only examined for participants in intervention arms (Early 1 and Early 2). 3 enrolled participants were assigned to groups (one participant to the 'Early 1' group and two participants to the 'Usual Care' group), but subsequently withdrawn from the study when it became clear that they did not meet eligibility criteria. As such, data for one 'Early 1' group participant was not included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 31 | 31 | 0
Participants | 7 | 6 | 0

5. Other Pre Specified Outcome: Enacted and Internalized Stigmas
Description: As measured by the HIV/AIDS Stigma Instrument-PLWA (HASI-P) Scale. The HASI-P is a 33-item scale that contains questions in 6 different stigma-related domains or factors. For each item, participants are asked to describe the frequency of experienced stigmatizing events in the past 3 months on a 4-point Likert scale (0- Never, 1- Once or twice, 2- Several times, or 3- Most of the time), with higher scores indicating greater stigma. The instrument is scored by summing the scores (0-3) for each item and then dividing by the number of items within each factor (enacted or internalized stigma).
Time Frame: Measured at 6 months after enrollment in ART care
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 30 | 31 | 24
score on a scale
  Enacted stigma | 1.00 (0.01) | 1.00 (0.00) | 1.02 (0.10)
  Internalized stigma | 1.35 (0.66) | 1.39 (0.80) | 1.27 (0.54)

6. Other Pre Specified Outcome: Participant Health-related Costs
Description: Repeated measures analysis of participant direct and indirect costs. While we initially planned to report measurements at 1-, 6- and 12-months after enrollment in ART care, we ultimately reported direct and indirect average costs at 12 months by adding the reported costs at each of the 3 time points to calculate the cost over the entire study period, and then dividing by the number of visits to the health center.
Time Frame: 12-months
Measure: Mean (Standard Deviation); unit: Rwandan Francs (currency)
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 30 | 31 | 24
Rwandan Francs (currency) | 4562 (4034) | 4817 (3716) | 4842 (3948)

7. Other Pre Specified Outcome: ART Adherence
Description: Repeated measures analysis of patient self-reported ART adherence
Time Frame: Measured at 12-months after enrollment in ART care
Measure: Mean (Standard Deviation); unit: Days of ART missed in last 30 days
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 30 | 31 | 24
Days of ART missed in last 30 days | 0.8 (1.2) | 1.1 (5.4) | 0.6 (1.1)

8. Other Pre Specified Outcome: ART Adherence
Description: Repeated measures analysis of patient self-reported ART adherence
Time Frame: Measured at 6 months after enrollment in ART care
Measure: Mean (Standard Deviation); unit: Days of ART missed in last 30 days
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 30 | 31 | 24
Days of ART missed in last 30 days | 0.9 (2.0) | 1.6 (5.5) | 0.6 (1.1)

9. Other Pre Specified Outcome: Perceived Quality of Life
Description: Repeated measures analysis of participant quality of life as measured by the EuroQOL-5 Dimension-5 Levels (EQ-5D-5L) Visual Analog Scale (VAS). The EQ-5D-5L is a 5-level scale that measures self-rated problems (no problems, slight problems, moderate problems, severe problems and extreme problems) in 5 domains (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) as well as self-rated health. For this measure, we chose to use only the VAS, which asks respondents to rate their overall health from 0-100, with higher scores indicating greater self-rated health.
Time Frame: Measured at 6 months after enrollment in ART care
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 30 | 31 | 24
score on a scale | 52.2 (11.5) | 53.6 (13.8) | 50.4 (14.6)

10. Other Pre Specified Outcome: Perceived Quality of Life
Description: as for outcome 9
Time Frame: Measured at 12 months after enrollment in ART care
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 30 | 31 | 24
score on a scale | 52.2 (10.3) | 54.5 (11.4) | 54.4 (10.1)

11. Other Pre Specified Outcome: Satisfaction With Care
Description: as for outcome 3
Time Frame: Measured at 6 months after enrollment in ART care
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 30 | 31 | 24
score on a scale
  Non-clinical | 3.96 (0.46) | 3.98 (0.26) | 4.04 (0.33)
  Clinical | 3.74 (0.18) | 3.72 (0.19) | 3.72 (0.21)

12. Other Pre Specified Outcome: Anticipated Stigma
Description: As measured by an adapted version of the HIV stigma scale (anticipated stigma). Anticipated stigma is rated on a 5-point Likert-type scale (Very Unlikely [1] to Very Likely [5]), with higher scores indicating greater stigma. Items are averaged to create a composite score.
Time Frame: Measured at 6 months after enrollment in ART care
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 30 | 31 | 24
score on a scale | 2.43 (0.57) | 2.37 (0.59) | 2.73 (0.66)

13. Other Pre Specified Outcome: Anticipated Stigma
Description: as for outcome 12
Time Frame: Measured at 12 months after enrollment in ART care
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 30 | 31 | 24
score on a scale | 2.41 (0.77) | 2.37 (0.52) | 2.45 (0.56)

14. Other Pre Specified Outcome: Enacted and Internalized Stigmas
Description: as for outcome 5
Time Frame: Measured at 12 months after enrollment in ART care
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early 1 | Early 2 | Usual Care
Number analyzed (Participants) | 30 | 31 | 24
score on a scale
  Enacted stigma | 1.00 (0.00) | 1.04 (0.20) | 1.05 (.018)
  Internalized stigma | 1.11 (0.40) | 1.21 (0.58) | 1.10 (0.27)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on participants during their participation in the study (12 months)
Arm/Group | Early 1 | Early 2 | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 2/28
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/28
Other Adverse Events (participants affected / at risk) | 3/31 | 1/31 | 2/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early 1 (N=31) | Early 2 (N=31) | Usual Care (N=28)
Became pregnant during study (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 1 (1)
Incarcerated during study (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Developed tuberculosis during study (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT04567693/Prot_SAP_001.pdf
  • Informed Consent Form (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT04567693/ICF_000.pdf